CLINICAL TRIAL: NCT07264790
Title: Assessment of Topical Minoxidil on Intraoperative Flap Perfusion and Cutaneous Flap Viability in Breast Reconstruction
Brief Title: Assessment of Topical Minoxidil on Intraoperative Flap Perfusion and Cutaneous Flap Viability in Breast Recon
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00116354
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Breast Reconstruction; Perfusion; Complications; High Risk for Breast Cancer; Genetic Predisposition
MeSH Terms: conditions — Genetic Predisposition to Disease | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minoxidil (Experimental): All participants in this study will receive two solutions at a pre-operative visit: study drug and placebo. Use of the solutions will be randomized which means participants will be instructed to apply one solution to one breast and the other solution to the other breast.
  Interventions: Drug: Minoxidil
- Hair mousse (Placebo Comparator): All participants in this study will receive two solutions at a pre-operative visit: study drug and placebo. Use of the solutions will be randomized which means participants will be instructed to apply one solution to one breast and the other solution to the other breast.
  Interventions: Drug: Hair mousse

INTERVENTIONS:
Drug: Minoxidil — Each participant will receive both topical agents in order to apply daily for 14-days prior to surgery.
  Arms: Minoxidil
Drug: Hair mousse — Each participant will receive both topical agents in order to apply daily for 14-days prior to surgery.
  Arms: Hair mousse

SUMMARY:
The purpose of the study is to determine whether pharmacologic delay using minoxidil in patients undergoing bilateral risk reducing mastectomy with reconstruction could achieve improvement in flap perfusion and flap viability at the time of surgery. Patients will undergo randomization of their breasts to determine which breast will receive the experimental intervention and which breast will serve as the internal control (receive placebo). The experimental breast will receive the novel pharmacologic delay treatment, 5% minoxidil, while the internal control breast will receive the current standard of care, which does not include any topical application prior to surgery - a placebo control will be used.

This will be a triple-blind study, where both the participants and investigators will be blinded to which breast will receive the intervention. The patients will receive two bottles "compound A" and "compound B" with directions from the pharmacy for which compound to apply to each breast.

Product will be applied for 2 weeks prior to planned surgery. Surgery will proceed without any changes to standard practice.

ELIGIBILITY:
Inclusion Criteria:

1. Female sex > 18 years old
2. Genetic predisposition to cancer
3. Undergoing bilateral prophylactic mastectomy with same-day breast reconstruction
4. Capable of giving informed consent

Exclusion Criteria:

1. Diagnosis of breast cancer
2. History of cancer
3. Currently pregnant or planning to be pregnant (for women of child-bearing potential)
4. Male sex

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — High-risk for breast cancer diagnosis with desire to proceed with breast reconstruction
Enrollment: 25 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility, as measured by recruitment rate | Day 1
  Rate of study participation from eligible patients undergoing bilateral risk-reducing mastectomy with tissue expander-based implant reconstruction
Feasibility, as measured by retention rate | 90 days
  Retention of enrolled participants until the clinical endpoint
Feasibility, as measured by rate of participant adherence to the protocol | 90 days
  Rate of adherence to the treatment protocol

SECONDARY OUTCOMES:
Flap perfusion, assessed by a blinded plastic surgeon | Day of surgery
  A third-party blinded plastic surgeon will visually evaluate flap perfusion, from preoperative and intraoperative photos, and SPY-QP video and use their clinical judgement to assess perfusion.
Flap perfusion, assessed by ICG angiography | Day of surgery
  Perfusion is assessed using "relative value," which quantifies fluorescence as a percentage (%) relative to a reference point.
Incidence of mastectomy skin flap necrosis | 90 days
Incidence of surgical complications | 90 days
Incidence of reoperations or definitive second-stage reconstruction | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Brett Phillips, MD, Principal Investigator — Duke University
Locations (1):
- Duke Health, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No